CLINICAL TRIAL: NCT03783871
Title: A Single-Arm, Prospective, Multicenter Study to Evaluate the Safety and Effectiveness of the NeuWave Certus Microwave Ablation System in Chinese Patients With Hepatocellular Carcinoma
Brief Title: NeuWave Microwave Ablation HCC China Study
Acronym: NW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ethicon, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEU_2017_07
Record Dates: First submitted 2018-11-30; First posted 2018-12-21 (Actual); Results first posted 2025-02-14 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Liver Tumor; Hepatocellular Carcinoma
Keywords: HCC
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Single-arm (Experimental): Subjects will be treated with microwave ablation.
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — Subjects will be treated with microwave ablation.

SUMMARY:
This is a single-arm, prospective, multicenter, study. Individuals who are assessed for microwave (MW) ablation of HCC in accordance with their institution's standard of care (SOC), who meet study entry criteria and sign the informed consent, will be enrolled. The patients will be treated with MW ablation and afterwards followed for up to 36 months after the original ablation procedure to assess efficacy and safety. In addition to the final analysis after all enrolled patients complete the 36-month observation period, a summary of selected endpoints will be provided after all enrolled patients have completed each of the 1-month and 12-month visits.

To provide sites with an opportunity to get equal experience in the use of the Certus system, there will 3 patients treated as part of a run-in phase. These patients will only be included in the safety set.

DETAILED DESCRIPTION:
Patients who have a single HCC tumor up to 5 cm or a maximum of 3 HCC tumors of up to 3 cm per tumor will receive the same procedure: microwave ablation using only the NeuWave Certus Microwave Ablation System. Patients in this study will come to their study site for the ablation procedure. After the ablation procedure, the patient will be observed, which in most cases is expected to be 2 to 3 hours, and afterwards may return home. If the Study Doctor decides it is warranted for patient safety, the patient will remain in the hospital longer.

A minimum of one MRI of the liver must be taken at Baseline/Screening to ascertain tumor type, location, and size. (Tumor size will be measured in longest diameter and the diameter that is perpendicular to this longest diameter; tumor size must be measured with at least 2D imaging.) Physicians who are experienced with tumor ablation will do all ablations percutaneously using only the NeuWave Certus Ablation System. During the ablation, patients will be under an anesthesia method as per the institution's SOC. Ultrasound and/or CT scan will be used to guide the probe to the tumor and confirm accurate placement of the probe prior to emitting the microwaves.

Within 7 days after ablation, contrast-enhanced MRI will be done to confirm the completion of the ablation procedure. According to the standard practice at each study site, ablation confirmation will be classified as:

* complete tumor ablation with adequate margin (A0).
* complete tumor ablation with insufficient margin (A1).
* incomplete tumor ablation (A2). Over the course of 3 years, patients will return to their study site for post ablation follow-up visits, which will be carried out per the Schedule of Activities (see Table 1 at the end of the Synopsis). The follow-up schedule will be based on the original ablation procedure date. A re-ablation for any reason will not re-start or change the follow-up visit schedule.

At every follow-up visit, every patient will be scanned with at least one MRI to see if there are any tumor foci at the edge of the ablation zone, which indicates tumor progression. Repeat microwave ablation (using the Certus Microwave Ablation System only) may be performed for recurrence of target tumor(s) or to achieve complete tumor ablation with adequate margin (A0) of the target tumor(s) if the initial ablation had an insufficient margin, if the treating physician deems appropriate and necessary.

While repeat ablations for a recurrence may be conducted at any point during the study duration, repeat ablations to correct an ablative margin may only be performed within the first 30 days of the original ablation (by Visit 3).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed primary or recurrent HCC determined in accordance with the institution's SOC procedure, a single tumor size up to 5 cm or a maximum of 3 tumors up to 3 cm per tumor. Tumor size must be measured with at least 2-dimensional (2D) imaging.
* Scheduled for microwave ablation of the liver.
* Performance status 0-2 (Eastern Cooperative Oncology Group classification).
* Functional hepatic reserve based on the Child-Pugh score (Class A or B).
* Give voluntary, written informed consent to participate in this study and willing to comply with study-related evaluation and procedure schedule.
* At least 18 years of age.

Exclusion Criteria:

1. ASA score ≥ 4.
2. Active bacterial or fungal infections which are clinically significantly.
3. Chemotherapy or radiation therapy for HCC performed within 30 days prior to the study procedure.
4. Patient with implantable pacemakers or other electronic implants.
5. Planned/ scheduled liver surgery.
6. Platelet count ≤ 50 × 109/L.
7. Patients with uncorrectable coagulopathy at time of screening based on investigator judgement. Severe blood coagulation dysfunction (bleeding tendency, prothrombin time [PT] was greater than normal control for 3~5 seconds, platelet count [PLT] was less than 50x109/L, and the international normalized ratio [INR] was greater than 1.5).
8. Patient with renal failure and on renal dialysis.
9. Scheduled concurrent procedure other than MW ablation in the liver.
10. Pregnant or breast feeding.
11. Physical or psychological condition which would impair study participation.
12. Participation in any other interventional clinical study within 1 month before screening and concurrently during the study.
13. The patient is judged unsuitable for study participation by the investigator for any other reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2024-01-17 (Actual); Study Completion 2024-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Leading PI; Jinhua Huang, Doctor, Principal Investigator — Co-PI; Xiaoyan Xie, Doctor, Principal Investigator — Co-PI; Bo Zhai, Doctor, Principal Investigator — CO-PI
Locations (4):
- China (4):
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - The First Affiliated Hospital，Sun Yat-sen University, Guangzhou, Guangdong
  - Chinese PLA General Hospital, Beijing
  - Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 143 participants signed the informed consent, 8 of whom were later screen failures as they did not meet all inclusion/exclusion criteria. These 8 participants were not treated with the NEUWAVE microwave ablation device.
Pre-assignment Details: 135 participants met all inclusion/exclusion criteria. All participants were treated with the NEUWAVE microwave ablation device. The first 3 participants at each of the 4 clinical sites (12 participants total) were part of the 'run-in' phase and the remaining 123 participants were part of the 'full-analysis set', used for statistical analysis.
Groups:
- Microwave Ablation With NEUWAVE: Each participant underwent microwave ablation with NEUWAVE for the treatment of a single HCC tumor up to 5 cm or up to three HCC tumors, no more than 3 cm per tumor, in accordance with the study protocol.
Period: Overall Study
Arm/Group | Microwave Ablation With NEUWAVE
Started | 135
Completed | 105
Not Completed | 30
Not completed — Withdrawal by Subject | 15
Not completed — Death | 13
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Participants who met all inclusion/exclusion criteria, were treated with the NEUWAVE microwave ablation device, and were not part of the 'run-in' phase.
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 123
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.6 (10.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 94
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 123
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 123
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Technical Efficacy
Description: Defined as a combination of A0 ablations (complete tumor ablation with a surrounding 5 mm margin) and A1 ablations ( complete tumor ablation with inadequate margins), based on contrast-enhanced MRI scans at 1 month (+/- 7 days) post-ablation.
Time Frame: Day 23 to Day 37
Population: Each participant underwent microwave ablation with NEUWAVE for the treatment of a single HCC tumor up to 5 cm or up to three HCC tumors, no more than 3 cm per tumor. This excludes the run-in participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 115
Participants | 107

2. Secondary Outcome: Technical Success
Description: Defined as the combination of A0 ablations (complete tumor ablation with a surrounding 5 mm margin) and A1 ablations (complete tumor ablation with inadequate margins) based on contrast-enhanced Magnetic Resonance Imaging (MRI) performed up to 7 days post-ablation.
Time Frame: Day 0 to Day 7
Population: Each participant underwent microwave ablation with NEUWAVE for the treatment of a single HCC tumor up to 5 cm or up to three HCC tumors, no more than 3 cm per tumor, in accordance with the study protocol. This excludes the run-in participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 119
Participants | 112

3. Secondary Outcome: Local Tumor Progression
Description: Local Tumor Progression (LTP) was the appearance of tumor foci at the edge of the ablation zone, after at least one contrast-enhanced follow-up MRI scan had documented adequate ablation and an absence of viable tissue in the target tumor and surrounding ablation margin by using imaging.
Time Frame: 1 Month to 36 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 123
Participants | 18

4. Secondary Outcome: Overall Survival
Description: Measured from the time of the initial ablation procedure to the time of death or last follow-up, if death has not occurred
Time Frame: 36 months
Population: Each participant underwent microwave ablation with NEUWAVE for the treatment of a single HCC tumor up to 5 cm or up to three HCC tumors, no more than 3 cm per tumor, in accordance with the study protocol. As this is a safety endpoint, it includes the run-in participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 135
Participants | 13

5. Secondary Outcome: Progression-Free Survival
Description: The length of time from the original ablation procedure until any type of disease progression (local, regional, or distant) or until death.
Time Frame: 36 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Microwave Ablation With NEUWAVE
Number analyzed (Participants) | 123
Participants | 81

ADVERSE EVENTS:
Time Frame: 36 Months
Description: Adverse Events (AEs) were defined as any undesirable clinical occurrence in a participant, whether attributable to the study device/procedure or not. AEs were captured for the first 30 days after the ablation procedure. After 30 days, only Serious Adverse Events (SAEs) were captured throughout the duration of the study (36 months).
Groups:
- Microwave Ablation With NEUWAVE: Each participant underwent microwave ablation with NEUWAVE for the treatment of a single HCC tumor up to 5 cm or up to three HCC tumors, no more than 3 cm per tumor, in accordance with the study protocol. Includes the run-in participants.
Arm/Group | Microwave Ablation With NEUWAVE
All-Cause Mortality (participants affected / at risk) | 13/135
Serious Adverse Events (participants affected / at risk) | 42/135
Other Adverse Events (participants affected / at risk) | 115/135
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation With NEUWAVE (N=135)
Gastroenteritis (Infections and infestations) | 3 (3)
Hepatic cirrhosis (Hepatobiliary disorders) | 7 (7)
Jaundice cholestatic (Hepatobiliary disorders) | 4 (5)
Cholecystitis (Hepatobiliary disorders) | 2 (2)
Hepatic function abnormal (Hepatobiliary disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (3)
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Biliary tract infection (Infections and infestations) | 2 (2)
Liver abscess (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Multiple organ dysfunction syndrome (General disorders) | 2 (2)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Esophageal varices hemorrhage (Gastrointestinal disorders) | 2 (2)
Myocardial infarction (Cardiac disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Microwave Ablation With NEUWAVE (N=135)
Hepatic function abnormal (Hepatobiliary disorders) | 66 (67)
Procedural pain (Injury, poisoning and procedural complications) | 43 (43)
C-reactive protein increased (Investigations) | 14 (14)
Serum amyloid A protein increased (Investigations) | 14 (14)
Pyrexia (General disorders) | 29 (29)
Hepatic cirrhosis (Hepatobiliary disorders) | 7 (7)
Incision site pain (Injury, poisoning and procedural complications) | 13 (13)
Abdominal pain upper (Gastrointestinal disorders) | 8 (9)
Neutrophil count increased (Investigations) | 12 (12)
Leukocytosis (Blood and lymphatic system disorders) | 10 (10)
Hypertension (Vascular disorders) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-06): https://cdn.clinicaltrials.gov/large-docs/71/NCT03783871/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/71/NCT03783871/SAP_001.pdf